CLINICAL TRIAL: NCT05361447
Title: Open Label Single Center Trial Evaluating the Efficacy and Safety of Diazepam in GAD65 Associated Epilepsy
Brief Title: Diazepam Trial in GAD65 Associated Epilepsy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study population was difficult to identify for enrollment interest.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kelsey M. Smith, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-007195
Record Dates: First submitted 2022-05-01; First posted 2022-05-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: GAD 65 Antibody-associated Epilepsy
MeSH Terms: interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GAD65 Associated Epilepsy (Experimental): Subjects diagnosed with GAD65 associated epilepsy, serum high-titer GAD65 positivity, trialed and failed at least 2 anti-seizure medications, at least 4 seizures per month will be started on diazepam.
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — 5 mg twice daily oral for 1 week and then increase to 10 mg twice daily oral
  Other Names: Valium

SUMMARY:
The purpose of this study is to determine whether diazepam reduces the frequency of seizures in GAD65 antibody associated epilepsy.

DETAILED DESCRIPTION:
GAD65 is an intracellular enzyme that plays a key role in the conversion of glutamate to gamma-aminobutyric acid (GABA), the primary inhibitory neurotransmitter in the CNS. Benzodiazepines augment the sensitivity of the GABA-A receptor to GABA, prolonging its inhibitory effect, perhaps enhancing the potential for neural inhibition in conditions in which GABA is depleted.

GAD65 antibodies have been identified in a subset of patients with drug resistant focal epilepsy and limbic encephalitis. While it has not been definitively determined that these antibodies cause GAD65 inhibition and GABA depletion directly, diazepam, a common benzodiazepine, has been established as a mainstay of therapy for stiffperson's syndrome, a condition that is commonly associated with GAD65 antibody positivity. Given these observations, diazepam has been used by the investigators in a small number of patients with intractable epilepsy in the setting of GAD65 antibody positivity, with some encouraging anecdotal results with one patient being rendered seizure free for three years.

The purpose of this study is to generate prospective data on use of diazepam in patients with epilepsy related to high-titer GAD65 antibody positivity.

ELIGIBILITY:
Inclusion Criteria:

* High-titer serum GAD65 positivity > 20 nmol/L High-titer serum GAD65 IgG seropositivity titer >20 nmol/L and/or CSF GAD65 seropositivity titer > 0.02 nmol/L.
* Drug-resistant focal epilepsy, having failed 2 previous anti-seizure medications.
* Stable treatment for the 1 month prior to enrollment.
* Patients must be able to give informed consent or have an appropriate representative available to do.

Exclusion Criteria:

* Alternative etiology for epilepsy.
* Already on another benzodiazepine.
* On a regularly scheduled opiate.
* Co-existing antibodies associated with seizures.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | Baseline, 3 months
  Median percentage change in the mean monthly frequency of seizures as measured by patient recorded seizure frequency

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Smith, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials